CLINICAL TRIAL: NCT06922513
Title: Clinical Feasibility of Mobile App-Based Self-Management for Breast Cancer-Related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JiHye Hwang, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SMC 2024-04-011; HA23C0423 (Other: National Cancer Center (NCC))
Record Dates: First submitted 2025-03-19; First posted 2025-04-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Related Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- digital health (Experimental): Unilateral Upper Limb Lymphedema Associated with Breast Cancer
  Interventions: Device: digital health (Application and Smart Measuring Tape)

INTERVENTIONS:
Device: digital health (Application and Smart Measuring Tape) — For lymphedema management, we use a smart measuring tape to measure arm circumference and provide analysis results along with self-management strategies.

SUMMARY:
The study evaluates a newly developed service that provides personalized self-management guidance based on evidence-based arm circumference measurements and resulting volume changes. The research aims to determine whether this digital solution is practical and acceptable for patients while identifying any unexpected challenges during implementation, ultimately establishing its potential for clinical integration into lymphedema care.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 70 years of age
* Diagnosed with breast cancer-related unilateral upper limb lymphedema
* Possessing an Android or iOS smartphone
* Voluntarily deciding to participate and providing written consent after receiving a detailed explanation of this study

Exclusion Criteria:

* Diagnosed with malignant lymphedema due to metastasis or recurrence
* Having severe comorbidities (underlying diseases, neuromusculoskeletal disorders, cognitive, mental, or visual impairments, etc.) that make it difficult to use the application and participate in exercise interventions

Discontinuation Criteria:

* Development of serious complications or cancer metastasis/recurrence during the study period
* Occurrence of a serious illness unrelated to study participation
* Failure to follow the instructions of the study physician
* Voluntary withdrawal from the study or development of circumstances preventing participation

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Usability and Acceptability | Baseline, Month 3
  Self-Developed Questionnaire A. One item on the necessity of a lymphedema self-management app B. 23 items on satisfaction and acceptability C. Scoring scale: 1 (Strongly Disagree) - 6 (Strongly Agree)
SUS | Baseline, Month 3
  Full Title: System Usability Scale A. A 10-item questionnaire to evaluate system usability B. Score range is 0-100, with a benchmark known to be 68 points Self-developed questionnaire

SECONDARY OUTCOMES:
TTM (Transtheoretical Model) | Baseline, Month 3
  Objective: behavior change stage Scoring System A. Assess health behavior change on a 5-step scale B. (1) Before consideration: No intention to change problem behavior or adopt healthy behavior within the next 6 months, (2) Consideration: No specific plan but plan to take action within the next 6 months, (3) Preparation: Plan to take action within the next 30 days, (4) Action: In progress (less than 6 months), (5) Maintenance: In progress (more than 6 months) C. Check whether the change in the stage has occurred in a positive direction
LYMQOL | Baseline, Month 3
  Full Title: Lymphedema quality of life questionnaire A. A questionnaire to measure the quality of life in patients with arm lymphedema B. Composed of subdomains including function, appearance, symptoms, mood, and quality of life C. Function, appearance, symptoms, and mood are rated on a 1-4 scale where lower scores indicate better quality of life, while quality of life is rated on a 0-10 scale where higher scores indicate better quality of life
EQ-5D-5L | Baseline, Month 3
  Full Title: EuroQol 5-Dimension 5-level Objective: quality of life Scoring System: Each item is evaluated on a 5-point scale and weighted according to the country. EQ VAS evaluates data on a scale of 0-100, with a higher score indicating better health.
self-efficacy | Baseline, Month 3
  Full Title: lymphedema-specific exercise barriers self-efficacy A. Composed of 9 general exercise barriers and 5 lymphedema-related barrier items B. Evaluates how confident one feels about exercising in each situation on a scale from 0% (not confident at all) to 100% (extremely confident) with 10% intervals C. Interpreted as '0-20%=not confident at all, 20-40%=slightly confident, 40-60%=moderately confident, 60-80%=very confident, 80-100%=extremely confident'
upper arm use | Baseline, Month 3
  Self-developed questionnaire A. Level of self-awareness of edema, amount of affected arm use, anxiety about using the affected arm B. Level of self-awareness of edema: 2 items, 0 (not at all) - 10 (very much) scale C. Amount of affected arm use: 1 item, change in arm usage on a -5 to 5 scale D. Anxiety about using the affected arm: 1 item, change in anxiety about arm use on a -5 to 5 scale
ICF (International Classification of Functioning, Disability, and Health) | Baseline, Month 3
  Objective: function, activity and participant, environment Scoring System: A. Assess the 8 items of body functions, 8 items of activities and participation, and 8 items of environmental factors of the breast cancer ICF core set brief B. Body functions are assessed as 0 (no problems) - 4 (extreme problems), 9 (not applicable). Activities and participation are assessed as 0 (no difficulties) - 4 (extreme difficulties), 9 (not applicable). Environment is assessed as 0 (no barriers) - 4 (extreme barriers), +0 (no facilitating factors) - +4 (complete facilitating factors), 9 (not applicable).
COPM | Baseline, Month 3
  Full Title: Canadian Occupational Performance Measure A. A client-centered assessment that identifies and prioritizes everyday problems that limit an individual's participation in daily life across all areas, including self-management, productive activities, and leisure B. Performance and satisfaction for activities selected as important issues are evaluated on a 0-10 scale C. Clinically significant change = 2-point change
Smart Measuring Tape | Baseline, Month 3
  Upper Limb Circumference Measurement
Perometer | Baseline, Month 3
  Optoelectronic Limb Volumeter (Perometer) Upper Limb Volume Measurement

OTHER OUTCOMES:
GPAQ | Baseline
  Full Title: Global Physical Activity Questionnaire Consists of 16 questions designed to estimate an individual's physical activity level and sedentary time across three domains (work, transportation, and leisure time)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Republic of Korea, South Korea

IPD SHARING:
Plan to Share IPD: No